CLINICAL TRIAL: NCT00999856
Title: Investigation of a Sub-Conjunctival Insert
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Two cohorts successfully completed; further cohorts not needed; no safety issue!
Sponsor: EyeSense GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Device Feasibility
Other Study IDs: P-2.1-C-01
Record Dates: First submitted 2009-09-28; First posted 2009-10-22 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Care
Keywords: medical device,; sub-conjunctival insert; photometer; fluorescence; subconjunctival interstitial fluid glucose; non-invasive measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Active Comparator): In the Cohort 1 an uncoated Insert and the photometer version 1 is used. Twelve trial subjects are appointed into 4 subgroups. The difference between these subgroups is the wearing time of the insert.
  Interventions: Device: GOMIS and Photometer
- Cohort 2 (Active Comparator): Cohort 2 consists of 12 trial subjects who are appointed to 2 subgroups. One group will wear the insert for a minimum of 12 month and the other group for a minimum duration of 18 month. In Cohort 2 an improved insert is used. The photometer will be the same than in cohort 1.
  Interventions: Device: GOMIS and Photometer
- Cohort 3 (Active Comparator): Cohort 3 only differs in the used photometer from cohort 2.
  Interventions: Device: GOMIS and Photometer
- Cohort 4 (Active Comparator): Twelve trial subjects are appointed to two subgroups that differ in the minimum wearing duration of the insert (12 month and 18 month). In Cohort 4 a new insert will be tested together with a better photometer.
  Interventions: Device: GOMIS and Photometer
- Cohort 5 (Active Comparator): The difference between Cohort 5 and Cohort 4 is that the best tested insert and the best evaluated photometer will be used.
  Interventions: Device: GOMIS and Photometer

INTERVENTIONS:
Device: GOMIS and Photometer — Insert is placed under the conjunctiva. During measurement sessions photometer will be placed in front of the eye in which the insert is located to perform the fluorescence measuring.
  Other Names: Ocular Mini Insert (OMI)
  Arms: Cohort 1
Device: GOMIS and Photometer — An improved insert is placed under the conjunctiva. During measurement sessions photometer will be placed in front of the eye in which the insert is located to perform the fluorescence measuring.
  Other Names: Ocular Mini Insert (OMI)
  Arms: Cohort 2
Device: GOMIS and Photometer — Insert is placed under the conjunctiva. During measurement sessions photometer version 2 will be placed in front of the eye in which the insert is located to perform the fluorescence measuring.
  Other Names: Ocular Mini Insert (OMI)
  Arms: Cohort 3
Device: GOMIS and Photometer — After comparing Photometer Version 1 and Version 2 the better one of them will be used for measurements in Cohort 4. A new insert will be implanted under the conjunctiva.
  Other Names: Ocular Mini Insert (OMI)
  Arms: Cohort 4
Device: GOMIS and Photometer — The insert version with the best results will be implanted. The photometer that was used in Cohort 4 will be taken again for fluorescence measurements.
  Other Names: Ocular Mini Insert (OMI)
  Arms: Cohort 5

SUMMARY:
The study is intended to evaluate a non-invasive method of glucose measurement in diabetics. The medical device that is evaluated consists on a sensor-insert which is placed under the conjunctiva of the eye of diabetic patients and a photometer. The goal is to prove that the sensor signal correlates with the blood glucose of the patients determined by standard laboratory blood glucose measurement.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age
* Insulin dependent diabetes requiring daily finger pricking to monitor blood glucose
* Sign written Informed Consent

Exclusion Criteria:

* Inability to follow the protocol schedule
* Participating in another clinical study
* Pregnant or lactating females
* Any ongoing condition that would prevent from proper handling of the instrument (e.g. blindness, strong impaired vision, impaired motor skills)
* Any known hypersensitivity to any of the products to be used in the study, including preservatives etc.
* Malignancies requiring therapy during the study
* Severe chronic diseases e.g. renal failure, liver cirrhosis etc. which may interfere with the conduct or completion of the study
* Poorly controlled diabetes mellitus with prior hemoglobin A1C greater than 10%
* Any ocular disease requiring topical medication besides those permitted by this protocol.
* Ocular or other condition which increase the risk of ocular surgery, e.g. acute or chronic conjunctivitis or blepharitis, corneal disorders, previous eye surgery or eye surgery within the following 12 weeks, coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2012-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
short term and mid term performance of different versions of the insert | at 1 month, at 2 months, at 3 months
recovery from surgery (wound healing) | at 1 month, at 2 months, at 3 months
demonstrate correlation between the fluorescence reading of the insert and capillary blood glucose measurement | at 1 month, at 2 months, at 3 months

SECONDARY OUTCOMES:
subjective impressions | 1 year
lag time between blood glucose and interstitial fluid glucose | at 1 month, at 2 months, at 3 months
signal to noise ration, signal drift and stability of measurement | at 1 month, at 2 months, at 3 months
conjunctival hyperemia | at 1 month, at 2 months, at 3 months
duty of care | at 1 month, at 2 months, at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hasslacher, Prof. Dr. med., Principal Investigator — Diabetes Institut Heidelberg, Germany; Gerd Auffarth, Prof. Dr. med., Principal Investigator — University Hospital Heidelberg, Ophthalmology, Heidelberg, Germany
Locations (1):
- Diabetes Instiut Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Hasslacher C, Auffarth G, Platten I, Rabsilber T, Smith B, Kulozik F, Knuth M, Nikolaus K, Muller A. Safety and accuracy of a new long-term subconjunctival glucose sensor. J Diabetes. 2012 Sep;4(3):291-6. doi: 10.1111/j.1753-0407.2012.00192.x. PMID 22341132
- See also: Publication of Study Data — http://www.ncbi.nlm.nih.gov/pubmed/22341132
- See also: EyeSense GmbH — http://www.eyesense.com/